CLINICAL TRIAL: NCT03897777
Title: Effects of Exercise on Hypertension and Gut Dysbiosis in African Americans
Brief Title: Exercise, Hypertension, and Gut Dysbiosis in African Americans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina Agriculture & Technical State University (Other)
Responsible Party: Principal Investigator, Marc D Cook, Assistant Professor of Exercise Immunology, North Carolina Agriculture & Technical State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NCarolinaATSU
Record Dates: First submitted 2019-01-26; First posted 2019-04-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hypertension
Keywords: Blood pressure; Gut dysbiosis; Exercise training
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypertension (Exercise Intervention) (Experimental): Participants with hypertension will submit blood and fecal samples for comparison to control participants with normal blood pressure. Control group will only donate fecal and blood samples and will not participate in the exercise intervention. Participants with hypertension will also perform 3 months of supervised aerobic exercise (5 days/week) and submit blood and fecal samples every 4 weeks until the completion of the study.
  Interventions: Behavioral: Exercise Training effect on Hypertension and Gut Dysbiosis

INTERVENTIONS:
Behavioral: Exercise Training effect on Hypertension and Gut Dysbiosis — the proposed research will: 1) Characterize gut microbial community structure in AA with hypertension in two important compartments that make up the overall gut bacteria in the colon (fecal and colon mucosa); 2) Quantify the relationship between aerobic exercise training and gut bacteria to identify SCFA microbes that adapt to exercise and benefit BP.

SUMMARY:
African Americans have the greatest burden of endothelial dysfunction and hypertension. Recently, gut microbial dysbiosis (a term that describes a poorly diverse gut microbial profile and lower short-chain fatty acid (SCFA) production) has been linked to hypertension and may be involved in the pathogenesis of hypertension in African Americans. African Americans have been reported to have lower gut SCFA and SCFA can reduce blood pressure. Exercise reduces blood pressure and improves gut dysbiosis (increases SCFA) and likely couples' improvements in gut microbial health and vascular function to reduce blood pressure. Thus, the goals of this research are to fill a critical void concerning the interaction of gut dysbiosis, hypertension, and utilizing exercise to identify gut microbial adaptations that accompany a reduction in blood pressure. The short-term implications of this work will advance the clinical communities understanding of the relationship between dysbiosis and the pathogenesis of hypertension in African Americans, while long term implications will promote identifying adaptable gut microbes associated with vascular health to aid in amending treatment strategies for hypertension.

DETAILED DESCRIPTION:
African Americans (AA) have the greatest burden of hypertension and elucidating the pathogenesis of this racial disparity is important for amending treatment strategies. Gut microbial dysbiosis has been linked to hypertension and has been characterized as low microbial composition of short chain fatty acid (SCFA) producing microbes. Reduced gut SCFA production has been observed in AA with disease, such as glucose intolerance and vitamin deficiency, and may be related to the pathogenesis of hypertension in this group. Preliminary data show that aerobic exercise improves the gut microbial profile and increases SCFA production in animal models and humans. Additional preliminary data show that the SCFA butyrate attenuates dysfunction in AA endothelial cells suggesting a role for SCFA in endothelial/vascular function. The proposed studies have been constructed to fill a critical void in our understanding of the pathogenesis of hypertension in AA involving the gut microbiome. The investigators hypothesize that lower SCFA production is associated with blood pressure in AA and exercise will be effective in reducing blood pressure by coupling improvements in gut microbial health (↑SCFA production) and vascular health. The proposed research will: 1) quantify the relationship between gut dysbiosis (reduced gut and circulating SCFA) and blood pressure in AA with hypertension and 2) quantify the impact of aerobic exercise training on gut microbial community structure, identify adaptable SCFA microbes related to blood pressure, blood concentrations of SCFA, and blood pressure in AA. The research will provide novel insight into the pathogenesis of hypertension, particularly in the health disparate AA population, and will facilitate the development of future mechanistic studies to advance the clinical communities understanding of the "gut-vascular axis" concerning endothelial function and vascular disease in AA.

ELIGIBILITY:
Inclusion Criteria

* Sedentary (regular aerobic exercise frequency ≤2 times per week and duration ≤20 minutes per session; sedentary profession);
* 30-50 years of age;
* Control normotensive (systolic BP: 90-120 mmHg/diastolic BP: 60-80 mmHg)
* Elevated to Stage 1 Hypertension (systolic BP: 120-129 mmHg/diastolic BP: 80-89 mmHg) and/or stage 1 hypertension (systolic BP: 130-159 mmHg/diastolic BP: 90-99 mmHg).

Exclusion Criteria

Diagnosed with any of the following:

* Uncontrolled hypertension, stroke, history of heart attack, heart disease;
* Metabolic disease (diabetes mellitus);
* Inflammatory diseases (inflammatory bowel disease(s), rheumatoid arthritis, and systemic lupus erythematosus);
* Kidney stones or gallbladder problems;
* Kidney disease;
* Liver disease;
* Lung disease;
* Cancer within the previous 6 months; (11) pregnant females;
* Peripheral vascular disease;
* Taking hypertension medications or those known to affect inflammation or metabolic function (anti-inflammatories, statins, thyroid medication) in the past 1 month;
* Currently smoking;
* Other conditions that would exclude vigorous exercise (>2mV ST-segment depression or CVD signs and symptoms during the screening graded exercise test).

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 3 months
  Expect a change in systolic and diastolic BP
Gut Dysbiosis | 3 months
  Expect an change in microbial diversity and SCFA producing microbes

CONTACTS AND LOCATIONS:
Overall Officials: Marc Cook, PhD, Principal Investigator — North Carolina Agriculture & Technical State University
Locations (1):
- North Carolina A&T State University, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identifiable IPD will be made available for all primary and secondary data measures.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available within 6 months of the end of the study

DOCUMENTS (1):
  • Informed Consent Form (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT03897777/ICF_001.pdf